CLINICAL TRIAL: NCT01317316
Title: Causes and Characteristics of Occupational Eye Injuries in Western Turkey
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Pamukkale University Medical Faculty, emergency department
Other Study IDs: Serinken 003
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2006-11

CONDITIONS: Other and Unspecified Superficial Injuries of Eye

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with work-related eye injuries (WREI) admitted to the center in the four-year period were enrolled in this prospective study. Institutional Review Board approval was obtained before commencement of the study. A special data recording system was developed for the study. The study sample comprised only the casualties occurred at workplace and while working de facto. The data were abstracted via face to face contact in the emergency department (ED). The data sheets comprised sociodemographic and injury-related information brought together in 15-item questionnaire. Causes of occupational injuries as reported by the victims were assigned to either of two groups: "Worker-related causes" and "workplace-related causes".

Since workers are known to be pressured by the workplace to work in unsafe ways, an isolated room in the ED was used for this purpose in order to prevent bias and the patients were not accompanied by any person other than the medical personnel in charge of due medical care. The patients were also assured that the information obtained by the survey are to be used for research purposes only and no feedback is to be given to employers or related persons.

Patients who did not give consent for the study, fatal accidents and patients younger than 15 years of age were excluded from the analysis.

DETAILED DESCRIPTION:
All data obtained in the study were recorded in and analyzed using the Statistical Package for Social Sciences for Windows, Version 17. Numerical variables were given as mean and standard deviation (SD), while categorical variables were given as frequencies (n) and percentages.

ELIGIBILITY:
Inclusion Criteria:

* The study sample comprised only the casualties occurred at workplace and while working de facto

Exclusion Criteria:

* Other

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with WREI admitted to the center in the four-year period were enrolled in this prospective study. Institutional Review Board approval was obtained before commencement of the study. A special data recording system was developed for the study. The study sample comprised only the casualties occurred at workplace and while working de facto.
Sampling Method: Non-Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2007-01; Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: mustafa serinken, MD, Study Director — Pamukkale University